CLINICAL TRIAL: NCT01034566
Title: Proton Radiotherapy for Retroperitoneal Sarcoma
Brief Title: Proton Beam Radiation Therapy in Treating Patients With Retroperitoneal Sarcoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to accrue
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 04509
Record Dates: First submitted 2009-12-04; First posted 2009-12-17 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Proton Therapy

STUDY DESIGN:
Intervention Model Description: Proton radiation for retroperitoneal sarcoma
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients undergo proton beam radiotherapy 5 days a week for 6 (preoperative patients) or 8 (post-operative patients) weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Proton Beam Radiation Therapy

INTERVENTIONS:
Radiation: Proton Beam Radiation Therapy

SUMMARY:
RATIONALE: Specialized radiation therapy, such as proton beam radiation therapy, that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue in patients with retroperitoneal sarcoma. PURPOSE: This phase I trial is studying the side effects and and best dose of proton beam radiation therapy in treating patients with retroperitoneal sarcoma.

DETAILED DESCRIPTION:
Detailed DescriptionPRIMARY OBJECTIVES:

I. To determine the feasibility and toxicity of proton radiotherapy for retroperitoneal sarcomas.

II. To determine the maximum safe proton radiotherapy dose for retroperitoneal sarcomas.

III. To determine the maximally tolerated dose of proton radiotherapy for patients with potentially resectable retroperitoneal sarcoma. (Pre-operative cohort) IV. To assess acute side effects from irradiation using proton beam therapy and dose/volume constraints that are derived from conventional radiotherapy. (Postoperative cohort)

SECONDARY OBJECTIVES:

I. To assess the clinical effectiveness of proton radiotherapy for retroperitoneal sarcoma.

II. To determine the long-term toxicity of proton radiotherapy to the abdomen and pelvis region.

III. To monitor for effects of proton treatment on tumor and normal tissues using radiographic imaging (both cohorts) or ex-vivo analysis of tissue samples (preoperative cohort only).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of sarcoma in the peritoneum/retroperitoneum/pelvis are eligible for this study
* Patients must have either radiographic(pre-operative) or pathologic (post-operative) evidence of disease limited the peritoneum/retroperitoneum/pelvis without evidence of peritoneal sarcomatosis
* For pre-operative cases, the patient must be considered operable/resectable as judged by the attending surgeon (this is determined by an extensive radiographic and medical evaluation that includes but is not limited to: CT Chest and Abdomen with contrast, MRI/CT Brain and Medical/Cardiac Clearance)
* Patients should have an EGOC status of 0-2
* Patients must sign a document that indicates that they are aware of the investigative nature of the treatment of this protocol, and the potential benefits and risks (patients unwilling or unable to sign informed consent are excluded from the study)
* Women of child-bearing potential as long as she agrees to use a recognized method of birth control (e.g. oral contraceptive, IUD, condoms or other barrier methods etc.); hysterectomy or menopause must be clinically documented

Exclusion Criteria:

* Prior or simultaneous malignancies within the past two years (other than cutaneous squamous or basal cell carcinoma, melanoma in situ or thyroid carcinoma)
* Pregnant women, women planning to become pregnant and women that are nursing
* Patients who experience surgical complications that prevent radiation from starting for 5 months or more, unless there is evidence of gross residual disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Acute toxicity as assessed by NCI CTC Version 3.0 | Within 60 days of completion of radiotherapy

SECONDARY OUTCOMES:
Late toxicity as assessed by the RTOG/EORTC late morbidity scoring system | After 60 days of therapy
Clinical efficacy | One year
  Local recurrence-free survival, distant metastasis-free survival, and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Curtiland Deville, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States